CLINICAL TRIAL: NCT05777200
Title: Sociodemographic and Clinical Characteristics of Patients Admitted to the Addiction Management Unit of Assiut University Hospital
Brief Title: Sociodemographic and Clinical Characteristics of Patients Admitted to the Addiction Management Unit
Status: Active, not recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mena Fahy Rizq Farag, Resident of Neurology and Psychiatry, Assiut University Hospital, Assiut University
Other Study IDs: Substance-use disorder
Record Dates: First submitted 2023-02-27; First posted 2023-03-21 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Substance Use Disorders
Keywords: substance use disorder; addiction; Sociodemographic characteristics; personality traits; patterns of substance abuse
MeSH Terms: conditions — Substance-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: Supportive psychotherapy — Counselling patients, providing supportive psychotherapy to help them detox their illicit drug usage, and help them rehabilitate again into society.

SUMMARY:
Substance use disorder (SUD) is a dynamic process that changes constantly over time with new trends of drug dependence emerge every now and then, thus timely information about trends in psychoactive substance use could yield tailored interventions and reduce potential harms.

Identifying personal, social, and demographic characteristics of patients with this disorder at the local, regional, and national levels helps physicians, health authorities, and policy-makers detect early emerging trends and enable them better plan and implement prevention, treatment, and rehabilitation programs.

This study aims to identify sociodemographic, personal characteristics, as well as patterns of illicit drug abuse in patients admitted for addiction treatment.

DETAILED DESCRIPTION:
Substance use disorder (SUD) is a complex condition in which there is uncontrolled use of a substance despite its harmful consequences. People with SUD have an intense focus on using a certain substance(s) such as alcohol, tobacco, or illicit drugs, to the point where the person's ability to function in day-to-day life becomes impaired. People keep using the substance even when they know it is causing or will cause problems.

Drug use brings with it the likelihood of several negative health consequences. These can include a wide range of physical and mental health disorders, foremost of which are dependence, HIV infection, hepatitis-related liver diseases, overdose and premature death.

The problem of substance use is becoming one of the most serious and rapidly growing phenomena all over the world. It accounts for substantial global morbidity, mortality, and financial and social burden. According to Global Burden of Disease (GBD) study, there were an estimated 494,000 drug-related deaths attributable to the use of drugs in 2019.

In 2020, 1 in every 18 people aged 15-64 worldwide - an estimated 284 million people (5.6 per cent of the population) - had used a drug in the past 12 months. However, the coverage of interventions for the treatment of drug use disorders remains low overall. Implementation of scientific evidence-based drug prevention interventions remains low as well, especially in middle- and low-income countries.

In Egypt, SUD is a serious public health threat. Recent studies have demonstrated increases in the prevalence of the use of tobacco, illegal drugs, and over-the-counter drugs, particularly among youth.

Drug treatment registers are often used as a proxy indicator of treatment demand. This information is useful for analysis of service utilization and can be used as an indicator of trends in prevalence and patterns of high-risk drug consumption.

Assiut University Hospital is the biggest hospital in Upper Egypt, and it provides health services for Assiut city and most of the neighboring governorates. Addiction management unit of Assiut University Hospital contains 16 beds, based on paid service and about 400 patients have been admitted per year.

SUD is a dynamic process that changes constantly over time with new trends of drug dependence emerge every now and then, thus timely information about trends in psychoactive substance use could yield tailored interventions and reduce potential harms.

Identifying personal, social, and demographic characteristics of patients with this disorder at the local, regional, and national levels helps physicians, health authorities, and policy-makers detect early emerging trends and enable them better plan and implement prevention, treatment, and rehabilitation programs.

This study aims to identify sociodemographic, personal characteristics, as well as patterns of illicit drug abuse in patients admitted for addiction treatment.

ELIGIBILITY:
Inclusion Criteria:

* All patients with substance use disorder who are admitted to the addiction treatment unit.
* Accept participating into the study.

Exclusion Criteria:

* Patients refuse participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with substance use disorder, based on DSM-5 criteria, who are admitted to the addiction management unit of Assiut University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-11-10 (Estimated)

PRIMARY OUTCOMES:
To identify the sociodemographic characteristics of patients with substance use disorder attending addiction treatment unit. | One week
  1. Sociodemographic characteristics with a special prepared survey that includes:
     * Personal information, and socioeconomic status.(Age, gender, marital status, work, income, educational level, ...etc)
     * Previous admissions/trials for detox.(number of previous admissions/trials detox, where they were, maximum abstinence time, and the withdrawal symptoms the patient had)
     * Medical, psychological, social, financial, and legal aspects of addiction.
     * Adverse life events dating before starting addiction.
     * Detailed description of substance(s) used.( Substances used, doses, route of administration, when, where, and with whom he prefers taking the drug)
  2. Psychiatric interview.
To identify personality traits of patients with substance use disorder attending addiction treatment unit. | One week
  Data about personality traits of patients with substance use disorder will be obtained through:
  1. Psychiatric interview.
  2. The Symptom Checklist-90-Revised (SCL-90-R).
  3. The Structured Interview for the Five-Factor Model of Personality (SIFFM).
  4. Addiction severity Index (ASI).
To identify patterns of substance abuse among patients with substance use disorder attending addiction treatment unit. | One week
  Data about patterns of substance abuse will be gathered through:
  1. Psychiatric interview.
  2. Addiction Severity Index (ASI).
  3. Urine Drug Screen.

CONTACTS AND LOCATIONS:
Overall Officials: Alaa El Din M. Darweesh, Prof., Study Chair — Department of Neurology and Psychiatry, Faculty of Medicine, Assiut University; Romany H. Gabra, Dr, Study Director — Department of Neurology and Psychiatry, Faculty of Medicine, Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Assiut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Loffredo CA, Boulos DN, Saleh DA, Jillson IA, Garas M, Loza N, Samuel P, Shaker YE, Ostrowski MJ, Amr S. Substance use by Egyptian youth: current patterns and potential avenues for prevention. Subst Use Misuse. 2015 Apr;50(5):609-18. doi: 10.3109/10826084.2014.997391. Epub 2015 Jan 28. PMID 25629955
- [Background] Connery HS, McHugh RK, Reilly M, Shin S, Greenfield SF. Substance Use Disorders in Global Mental Health Delivery: Epidemiology, Treatment Gap, and Implementation of Evidence-Based Treatments. Harv Rev Psychiatry. 2020 Sep/Oct;28(5):316-327. doi: 10.1097/HRP.0000000000000271. PMID 32925514
- [Background] Darweesh, A. E., Agban, M., Mohammed, M. H., & Gabra, R. H. (2020). Association between opioid use disorder (tramadol) and serum level of interleukin-2. Middle East Current Psychiatry, 27(1). https://doi.org/10.1186/s43045-020-00037-w
- [Background] Rabie, M., Shaker, N.M., Gaber, E. et al. Prevalence updates of substance use among Egyptian adolescents. Middle East Curr Psychiatry 27, 4 (2020). https://doi.org/10.1186/s43045-019-0013-8
- See also: Global Burden of Disease (2019) study. (n.d.). GBD results. Institute for Health Metrics and Evaluation. Retrieved September 23, 2022 — https://vizhub.healthdata.org/gbd-results
- See also: American Psychiatric Association. (n.d.). What is a substance use disorder? Psychiatry.org - What Is a Substance Use Disorder? Retrieved September 23, 2022 — https://psychiatry.org/patients-families/addiction-substance-use-disorders/what-is-a-substance-use-disorder